CLINICAL TRIAL: NCT01178242
Title: Salivary Gland and Labial Mucous Membrane Transplantation in the Treatment of Severe Symblepharon and Dry Eye in Patients With Stevens-Johnson Syndrome.
Brief Title: Salivary Gland Transplantation in the Treatment of Dry Eye in Patients With Stevens-Johnson Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Ana Estela Besteti Pires Ponce Santa Anna, MD, PhD, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0427/08
Record Dates: First submitted 2010-01-19; First posted 2010-08-10 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Symblepharon; Dry Eye; Ocular Surface Disease; Transplantation
Keywords: Labial mucous membrane; symblepharon; dry eye; Stevens -Johnson syndrome; salivary gland; ocular surface disease; transplantation
MeSH Terms: conditions — Dry Eye Syndromes; Stevens-Johnson Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Salivary Gland and Labial Mucous Membrane Transplantation (Experimental)
  Interventions: Procedure: Salivary Gland and Labial Mucous Membrane Transplantation

INTERVENTIONS:
Procedure: Salivary Gland and Labial Mucous Membrane Transplantation — Minor salivary glands (SG) will be obtain "en block" from the same donor site, at the inferior or superior labial mucous membrane, above the orbicularis oris muscle to correct lubrication. The thin split thickness graft of mucous membrane will be suture to the sclera with absorbable sutures

SUMMARY:
The purpose of this study is to evaluate salivary gland and labial mucous membrane transplantation in patients with severe symblepharon and dry eye secondary to Stevens-Johnson Syndrome (SJS).

DETAILED DESCRIPTION:
This study was performed to evaluate the use of salivary gland and labial mucous membrane transplantation in patients with severe symblepharon and dry eye secondary to SJS. Labial mucous membrane and salivary gland transplantation showed to be a good option in the treatment of severe symblepharon and dry eye secondary to SJS. labial mucous membrane, salivary glands, symblepharon, entropion, transplantation, graft.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with poor visual acuity, less or equal to 20/200, and Schirmer I test equal to zero.
* Eyes with symblepharon or ankyloblepharon that did not allow the placement of a Schirmer test strip will be consider not measurable.

Exclusion Criteria:

* Active infection and corneal melting or perforation.

Ages: 10 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
A Complete ophthalmic exam including Schirmer I test , slit lamp exam, fundoscopy will be perform before and six months after surgery. Symptons improvement considered positive if patients will refer improvement of eye moisturasing and motility. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- UNIFESP, São Paulo, São Paulo, Brazil